CLINICAL TRIAL: NCT06496386
Title: Robotic Assisted Major Lung Resection in Elderly Patients: Results From a Retrospective Study
Brief Title: Robotic Assisted Major Lung Resection in Elderly Patients
Acronym: ELDERLY
Status: Recruiting | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Pierluigi Novellis, Medical doctor, Scientific Institute San Raffaele
Other Study IDs: CET 234-2024
Record Dates: First submitted 2024-06-28; First posted 2024-07-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
Keywords: robot-assisted thoracoscopic surgery; lung resection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- very elderly patients: patients older than 80 years
- elderly patients: patients younger than 80 years

SUMMARY:
The study is a retrospective observational study. The study is designed to be multicentric and it will analyze medical records from selected patients that underwent major lung resection using DaVinci surgical platform performed in the participating centers.

There are no risks for the patients, as this is a retrospective data collection.

DETAILED DESCRIPTION:
The investigators will recruit all patients who underwent major lung resection (segmentectomy, lobectomy, bilobectomy, or pneumonectomy using a robotic system) from May 2015 to December 2022.

Patients are divided into two groups: older than 80 years (case- very elderly patients) and younger than 80 years (control- elderly).

the aim: Minimally invasive techniques such as robot-assisted thoracoscopic surgery (RATS) can potentially reduce surgical trauma and therefore prove particularly beneficial for elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years at the moment of surgery
* Suspected or confirmed diagnosis of lung cancer
* The patient can be candidate in terms of cardiac, kidney, liver and respiratory function the primary pathology is under control or controllable
* Absence of extrapulmonary metastases that are not controlled or controllable
* All procedures included use of DaVinci robot system

Exclusion Criteria:

* Age < 18 years at the moment of surgery
* Patients who cannot undergo surgery, as they do not meet the conditions outlined above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study will focus on the population of subjects undergoing lung resection with the DaVinci surgical platform from May 2015 to December 2022.
  The anatomical resections considered will be segmentectomy, lobectomy, bilobectomy or pneumonectomy using robotic system.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The perioperative complications | from the surgery at 30-90 days after
  the investigators will measure the perioperative complications of robotic lung resection in patients with 80 or more than 80 years (very elderly patients) compared to those with less than 80 years. Complications will be categorized according to the Clavien-Dindo scale.
spirometry tests | from hospitalizzation to the discharge date at maximum one week
  the investigators will measure the pre-operative respiratory function (Forced expiratory volume (FEV) , forced vital capacity (FVC)), in the two groups .
Postoperative hospital stay | from hospitalizzation to the discharge date at maximum one week
  the investigators will measure the post-operative hospital stay in days in the two groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Scientific Institute Ospedale San Raffaele, Milan